CLINICAL TRIAL: NCT02798978
Title: A 2-part Randomized, Double-blind (Sponsor-unblinded), Placebo-controlled, Ascending Dose and Parallel Group Study of TLR4 Agonist (GSK1795091) Administered to Healthy Subjects
Brief Title: A Phase I, 2-part (Part 1 Being a Single Dose Escalation and Part 2, a Parallel Group) Study of Toll-like Receptor (TLR4) Agonist (GSK1795091) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204685; 2016-000759-28 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Neoplasms
Keywords: pharmacokinetics; TLR4 agonist; cancer; tolerability; GSK1795091; pharmacodynamics; safety
MeSH Terms: conditions — Neoplasms | interventions — TLR4 agonist GSK1795091

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: GSK1795091 or Placebo (Experimental): In Part 1, subjects in sequential cohorts will receive single ascending doses of intravenous (IV) injection of GSK1795091 or matching placebo, with a starting dose of 7 nanogram (ng), on Day 1 until the highest dose is evaluated.
  Interventions: Drug: GSK1795091; Drug: Placebo
- Part 2 Cohort 1: GSK1795091 (Experimental): In Part 2 Cohort 1, subjects will receive IV injection of GSK1795091 on Day 1, at dose determined in part 1, and second dose on Day 8 (one week apart)
  Interventions: Drug: GSK1795091
- Part 2 Cohort 2: GSK1795091 (Experimental): In Part 2 Cohort 2, subjects will receive IV injection of GSK1795091 on Day 1, at dose determined in part 1, and a second dose on Day 15 (two weeks apart)
  Interventions: Drug: GSK1795091

INTERVENTIONS:
Drug: GSK1795091 — GSK1795091 will be supplied as solution for injection vial. Each 5 mL vial contains 0.001 milligram/mL (mg/mL; 1000 ng/mL) or 0.0001 mg/mL (100 ng/mL)of GSK1795091 and will be administered as IV bolus over 2-5 minutes (min) followed by a IV bolus of 10 mL normal saline.
Drug: Placebo — Matching placebo will be supplied as a solution for injection vial and will be administered as IV bolus over 2-5 min followed by a IV bolus of 10 mL normal saline
  Arms: Part 1: GSK1795091 or Placebo

SUMMARY:
This study is an ascending dose first-time-in-human study to determine the safety, tolerability, pharmacodynamic (PD), and pharmacokinetics (PK) profile of GSK1795091 in healthy subjects. The results will support the design of future clinical trials of GSK1795091 administered to subjects with advanced malignancies in combination with immune system modulators.

Part 1 will be a randomized, double-blind (sponsor-unblinded), placebo-controlled, single center, single dose escalation, sequential group evaluation of intravenously administered GSK1795091 to evaluate the safety and tolerability in healthy subjects. Part 2 will be an open-label, parallel group evaluation of 2 doses of GSK1795091 administered, either 1 week apart (Part 2, Cohort 1) or 2 weeks apart (Part 2, Cohort 2). In Part 2, on Day 1, subjects will receive intravenous GSK1795091 at a dose determined by results from Part 1. The total duration of this study is approximately 10 weeks from screening to the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs and 12-lead ECG. (A subject with a clinically insignificant abnormality or laboratory parameter(s) may be included only if the Investigator documents that the finding is unlikely to represent a safety risk and will not interfere with the study procedures.)
* Body weight 55-95 kilogram (kg) and body mass index within the range 19-30 kg/meter (m)^2 (inclusive).
* Male or Female of non-childbearing potential:

Males: Male subjects with female partners of child bearing potential must comply with the pre specified contraception requirements.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotropin test), not lactating, and is either of non-reproductive potential or reproductive potential. If of reproductive potential, then the subject should agree to follow one of the options listed per GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential from 30 days prior to the first dose and until 30 days after the last dose of study medication The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception

* Capable of giving signed informed consent

Exclusion Criteria:

* History of any significant medical condition (e.g. cardiac, pulmonary, metabolic, renal, gastrointestinal, rheumatological, etc.)
* History of frequent (>1 per week) headache or myalgia, asthma, syncope.
* History of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* Alanine aminotransferase (ALT) and bilirubin >1.1×upper limit of normal (ULN; isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Vital signs:

Systolic blood pressure (SBP) <90 and >140 milliliter of mercury (mmHg); diastolic BP <50 and >90 mmHg; heart rate (HR) <50 and >90 beats per minute (bpm); temperature >37.5 degree Celsius

* Clinically significant ECG abnormality and/or HR < 50 and >90 bpm; PR interval >220 milliseconds (msec); QRS duration >120 msec; and QTcF > 450 msec
* Anticipated requirement for any prescription medication during the study
* History of regular alcohol consumption within 6 months of the study averaging a weekly intake of >14 drinks for males or >7 drinks for females or inability to abstain from alcohol from 1 day prior to the inpatient period of the study until discharge (one drink is equivalent to 8 grams of alcohol: 200 milliliter [mL] of beer, 100 mL of wine or 1 measure (25 mL) of spirits)
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 2 months prior to screening or inability to abstain from smoking during the study
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Presence of hepatitis B surface antigen, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid polymerase chain reaction test is obtained.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency antivirus antibody.
* Donation of blood or blood products in excess of 500 mL within a 56-day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first visit (Day -2) in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first visit (Day -2).
* Exposure to GSK1795091 in a previous cohort of this study.
* Subject is unable to refrain from taking non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Subject is able to understand and communicate in German/or native language of the site. Subject, or close relative of the subject, is the investigator or a sub-investigator, research assistant, pharmacist, study coordinator, or other staff directly involved with the conduct of the study at that site
* Vulnerable subjects (eg subjects kept in detention)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20725

REFERENCES:
- [Background] Hug BA, Matheny CJ, Burns O, Struemper H, Wang X, Washburn ML. Safety, Pharmacokinetics, and Pharmacodynamics of the TLR4 Agonist GSK1795091 in Healthy Individuals: Results from a Randomized, Double-blind, Placebo-controlled, Ascending Dose Study. Clin Ther. 2020 Aug;42(8):1519-1534.e33. doi: 10.1016/j.clinthera.2020.05.022. Epub 2020 Jul 30. PMID 32739049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to be conducted in 2-parts, however Part 2 was discontinued by the Sponsor prior to its scheduled start. Part 1 was single-dose escalation, sequential group evaluation of intravenously administered GSK1795091 to evaluate the safety and tolerability in healthy participants.
Pre-assignment Details: Forty two participants were randomized in Part 1 of which 2 did not receive dose due to abnormal findings during pre-dose examination. Participants were randomized in ratio of 3:1 to receive GSK1795091 or matching placebo.
Groups:
- Part 1: Placebo: Participants in Part 1 were randomized to receive intravenous (IV) matching Placebo of GSK1795091. Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 7 ng: In Part one sequential group evaluation, participants were randomized to receive single IV dose of GSK1795091 7 nanogram (ng). Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 21 ng: In Part one sequential group evaluation, participants were randomized to receive single IV dose of GSK1795091 21 ng. Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 60 ng: In Part one sequential group evaluation, participants were randomized to receive single IV dose of GSK1795091 60 ng. Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 Repeated 60 ng: In Part one sequential group evaluation, participants were randomized to receive single IV repeat dose of GSK1795091 60 ng as the study was restarted. Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 100 ng: In Part one sequential group evaluation, participants were randomized to receive single IV dose of GSK1795091 100 ng. Participants were observed inpatient until discharge on Day 5.
- All Participants in Part 2: In part 2, two doses GSK1795091 determined by results from Part 1 were planned in parallel group evaluation. Part 2 was discontinued by the Sponsor prior to its scheduled start and no participants were enrolled.
Period: Part 1 (30 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng | All Participants in Part 2
Started | 10 | 6 | 6 | 6 | 6 | 6 | 0
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (45 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng | All Participants in Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 was discontinued by the Sponsor prior to its scheduled start.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng | All Participants in Part 2 | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 0 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.2 (8.42) | 30.2 (6.62) | 40.5 (7.64) | 39.7 (7.47) | 43.3 (8.43) | 38.3 (6.02) |  | 37.6 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 0 |  | 1
  Male | 10 | 6 | 6 | 6 | 5 | 6 |  | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Row 2: Black or African American | 1 | 0 | 0 | 0 | 1 | 0 |  | 2
  Row 2: White/Caucasian/European Heritage | 9 | 6 | 6 | 6 | 5 | 6 |  | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or events associated with liver injury and impaired liver function were categorized as SAE. All participants enrolled into the study who have received a dose of study medication (GSK1795091 or placebo) were included in the All Subjects Population. Participants with non-serious AEs (5 percentage threshold) and SAEs has been reported.
Time Frame: Up to Day 32
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo: Participants in Part 1 were randomized to receive IV matching Placebo of GSK1795091. Participants were observed inpatient until discharge on Day 5.
- Part 1: GSK1795091 7 ng: In Part one sequential group evaluation, participants were randomized to receive single IV dose of GSK1795091 7 ng. Participants were observed inpatient until discharge on Day 5.
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0
  Non-SAE (>= 5%) | 0 | 2 | 0 | 5 | 3 | 5

2. Primary Outcome: Change From Baseline in Body Temperature Part 1
Description: Body temperature was measured in semi-supine position after 5 minutes rest. Baseline values are the last non-missing pre-dose assessments. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value.
Time Frame: Baseline, Day 1 (1, 2, 4, 6, 8, 12, 16 hours), Day 2, Day 3, Day 4, Day 5, and Day 7.
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Celsius
  Day 1, 1 hour | 0.14 (0.084) | 0.17 (0.163) | 0.08 (0.264) | 0.15 (0.187) | 0.15 (0.281) | 0.17 (0.327)
  Day 1, 2 hour | 0.17 (0.095) | 0.23 (0.163) | 0.32 (0.232) | 0.68 (0.354) | 0.40 (0.179) | 0.87 (0.367)
  Day 1, 4 hour | 0.26 (0.196) | 0.42 (0.147) | 0.55 (0.389) | 0.98 (0.556) | 0.63 (0.383) | 1.25 (0.295)
  Day 1, 6 hour | 0.43 (0.206) | 0.53 (0.301) | 0.45 (0.464) | 0.82 (0.665) | 0.38 (0.483) | 0.93 (0.163)
  Day 1, 8 hour | 0.41 (0.197) | 0.53 (0.273) | 0.43 (0.301) | 0.63 (0.432) | 0.57 (0.258) | 0.75 (0.389)
  Day 1, 12 hour | 0.14 (0.255) | 0.18 (0.337) | 0.28 (0.397) | 0.28 (0.397) | 0.23 (0.242) | 0.67 (0.294)
  Day 1, 16 hour | 0.03 (0.258) | 0.02 (0.223) | -0.08 (0.319) | 0.03 (0.175) | 0.03 (0.225) | 0.32 (0.349)
  Day 2 | 0.06 (0.190) | -0.02 (0.172) | -0.05 (0.226) | 0.12 (0.147) | -0.08 (0.117) | 0.13 (0.186)
  Day 3 | -0.10 (0.221) | 0.07 (0.207) | -0.17 (0.225) | 0.10 (0.179) | -0.13 (0.250) | -0.08 (0.204)
  Day 4 | 0.01 (0.197) | 0.25 (0.259) | -0.15 (0.217) | 0.05 (0.266) | 0.02 (0.223) | -0.12 (0.204)
  Day 5 | 0.14 (0.178) | 0.22 (0.147) | -0.12 (0.194) | 0.17 (0.273) | -0.13 (0.250) | 0.13 (0.234)
  Day 7 | 0.02 (0.199) | 0.12 (0.204) | -0.13 (0.314) | 0.08 (0.354) | -0.20 (0.415) | 0.10 (0.228)

3. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) Part 1
Description: Systolic and diastolic BP was measured in semi-supine position after 5 minutes rest. Baseline values are the last non-missing pre-dose assessments. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value.
Time Frame: Baseline, Day 1 (1, 2, 4, 6, 8, 12, 16 hours), Day 2, Day 3, Day 4, Day 5, and Day 7.
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Millimeter of mercury (mmHg)
  DBP, Day 1, 1 hour | -2.1 (6.14) | -3.8 (2.79) | -2.3 (5.50) | -1.3 (4.27) | -3.2 (5.23) | -3.3 (4.18)
  DBP, Day 1, 2 hour | -4.3 (4.00) | -5.0 (1.26) | -5.0 (10.06) | -6.5 (2.43) | -4.8 (3.43) | -7.0 (8.20)
  DBP, Day 1, 4 hour | -1.9 (4.77) | -3.8 (3.54) | -3.7 (5.05) | -3.7 (5.82) | -4.5 (4.14) | -4.2 (4.88)
  DBP, Day 1, 6 hour | -0.5 (4.86) | -6.0 (4.86) | -3.5 (6.09) | -5.3 (8.21) | -0.8 (6.34) | -7.5 (6.38)
  DBP, Day 1, 8 hour | 0.9 (5.17) | -0.5 (2.95) | -2.3 (5.47) | -4.3 (10.73) | -0.8 (5.23) | -6.8 (6.85)
  DBP, Day 1, 12 hour | -2.2 (6.01) | -0.3 (6.25) | -2.7 (11.17) | -2.8 (5.27) | -4.3 (7.03) | -2.0 (8.32)
  DBP, Day 1, 16 hour | -3.2 (6.00) | -5.5 (8.87) | -5.8 (15.22) | -6.2 (5.88) | -3.8 (5.04) | -2.7 (10.13)
  DBP, Day 2 | 0.0 (5.40) | 1.0 (6.10) | -5.3 (8.80) | -1.0 (6.66) | 1.3 (7.87) | 0.7 (7.00)
  DBP, Day 3 | 0.1 (6.30) | -1.3 (5.39) | -5.0 (8.99) | 4.3 (10.89) | 1.0 (6.51) | 0.8 (7.08)
  DBP, Day 4 | 2.6 (9.38) | 0.7 (8.41) | -6.2 (11.29) | -2.2 (9.62) | -1.0 (4.10) | -1.0 (6.23)
  DBP, Day 5 | 2.4 (5.02) | 4.2 (4.54) | -1.2 (10.25) | 1.5 (10.45) | 1.5 (2.07) | 2.5 (6.06)
  DBP, Day 7 | 0.9 (7.03) | 3.7 (6.71) | -1.8 (7.86) | 4.7 (9.22) | 1.3 (6.31) | 3.2 (9.43)
  SBP, Day 1, 1 hour | 6.5 (5.78) | 4.7 (8.89) | 1.5 (9.05) | 8.8 (8.16) | 3.3 (6.12) | -1.3 (14.60)
  SBP, Day 1, 2 hour | -2.0 (6.53) | -1.2 (5.56) | -1.2 (11.23) | -3.7 (8.52) | 1.2 (7.08) | 0.8 (6.05)
  SBP, Day 1, 4 hour | -1.6 (4.25) | -1.0 (7.56) | -4.2 (11.99) | 0.3 (6.35) | 1.7 (8.55) | 1.2 (3.37)
  SBP, Day 1, 6 hour | 5.0 (8.65) | 4.2 (4.31) | 2.2 (11.70) | 1.8 (10.46) | 7.5 (9.35) | 3.2 (6.46)
  SBP, Day 1, 8 hour | 0.7 (8.04) | 2.3 (5.68) | 0.8 (17.78) | -2.7 (10.98) | 2.5 (6.25) | -2.3 (4.72)
  SBP, Day 1, 12 hour | 3.9 (11.56) | 2.3 (4.32) | 6.0 (19.76) | 6.2 (5.85) | 6.2 (9.68) | 2.0 (7.21)
  SBP, Day 1, 16 hour | -1.8 (6.16) | -6.8 (6.43) | -7.2 (22.51) | -6.8 (8.11) | -1.0 (14.10) | 0.8 (13.29)
  SBP, Day 2 | -3.2 (7.15) | -1.8 (3.60) | -5.0 (17.44) | -2.3 (11.54) | -0.7 (5.16) | 2.2 (6.85)
  SBP, Day 3 | -2.0 (10.09) | -1.3 (5.89) | -7.8 (15.94) | 5.0 (8.39) | 1.8 (5.12) | 1.0 (8.81)
  SBP, Day 4 | 0.7 (6.50) | -1.7 (8.38) | -8.2 (19.86) | -1.8 (12.88) | -1.7 (5.85) | -0.3 (2.66)
  SBP, Day 5 | 4.2 (4.69) | 1.5 (3.08) | -2.5 (17.76) | 9.5 (13.43) | 5.0 (4.65) | 4.0 (5.37)
  SBP, Day 7 | -0.1 (6.81) | 5.3 (8.91) | -4.3 (14.96) | 2.3 (10.78) | 1.5 (11.50) | 5.2 (7.83)

4. Primary Outcome: Change From Baseline in Pulse Rate Part 1
Description: Pulse rate was measured in semi-supine position after 5 minutes rest. Baseline values are the last non-missing pre-dose assessments. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value.
Time Frame: Baseline, Day 1 (1, 2, 4, 6, 8, 12, 16 hours), Day 2, Day 3, Day 4, Day 5, and Day 7.
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Beats per minute
  Day 1, 1 hour | 8.1 (6.92) | 8.2 (3.31) | 11.8 (7.65) | 16.7 (7.66) | 12.0 (5.10) | 10.2 (4.88)
  Day 1, 2 hour | 5.9 (5.36) | 8.2 (8.57) | 11.3 (11.74) | 17.5 (8.60) | 14.8 (9.45) | 14.3 (7.45)
  Day 1, 4 hour | 5.0 (7.67) | 2.8 (2.99) | 11.7 (15.12) | 17.8 (20.22) | 17.3 (9.79) | 20.8 (5.42)
  Day 1, 6 hour | 8.7 (6.73) | 8.7 (3.98) | 10.8 (13.12) | 15.7 (17.07) | 17.7 (7.37) | 15.7 (5.09)
  Day 1, 8 hour | 3.2 (6.49) | 1.7 (3.20) | 4.7 (6.15) | 4.7 (8.87) | 8.2 (5.74) | 6.3 (5.35)
  Day 1, 12 hour | 4.6 (8.45) | 4.7 (5.99) | 5.2 (15.48) | 7.2 (4.07) | 10.5 (4.59) | 9.0 (6.57)
  Day 1, 16 hour | -1.9 (5.55) | -2.0 (4.94) | -0.8 (19.77) | -0.7 (5.61) | 3.2 (2.64) | 2.8 (5.56)
  Day 2 | 0.3 (4.37) | -0.3 (3.78) | 1.0 (7.64) | 4.3 (6.12) | 0.5 (4.04) | 1.7 (8.16)
  Day 3 | 1.4 (3.27) | 5.5 (4.37) | -1.3 (12.71) | 7.0 (7.62) | 2.0 (3.16) | -1.2 (5.71)
  Day 4 | 3.2 (7.69) | 4.8 (7.60) | -1.3 (13.84) | 4.5 (4.97) | 2.2 (6.21) | -2.3 (3.83)
  Day 5 | 7.3 (8.58) | 6.3 (6.41) | 2.2 (14.69) | 4.5 (5.24) | 4.5 (7.56) | 2.7 (3.01)
  Day 7 | 7.4 (5.50) | 7.0 (4.43) | 1.7 (10.46) | 3.8 (7.19) | 6.7 (13.41) | 3.8 (5.19)

5. Primary Outcome: Change From Baseline in Respiratory Rate Part 1
Description: Respiratory rate was measured in semi-supine position after 5 minutes rest. Baseline values are the last non-missing pre-dose assessments. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value.
Time Frame: Baseline, Day 1 (1, 2, 4, 6, 8, 12, 16 hours), Day 2, Day 3, Day 4, Day 5, and Day 7.
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Breaths per minute
  Day 1, 1 hour | 0.2 (1.03) | 1.2 (0.41) | -0.2 (1.17) | 1.2 (2.93) | -0.2 (1.60) | -0.2 (1.94)
  Day 1, 2 hour | 0.3 (1.49) | 0.2 (0.75) | -0.2 (0.75) | 1.3 (3.08) | 1.0 (0.89) | 0.2 (1.94)
  Day 1, 4 hour | 0.2 (1.14) | 0.0 (1.79) | -0.2 (2.93) | 1.0 (2.00) | 1.2 (2.04) | 1.5 (4.04)
  Day 1, 6 hour | 0.9 (2.96) | 0.3 (2.34) | -0.7 (1.51) | -0.3 (2.34) | 1.5 (2.74) | 0.7 (3.27)
  Day 1, 8 hour | 1.3 (2.31) | 1.0 (2.68) | -0.3 (1.97) | 0.8 (4.36) | 0.8 (1.72) | -0.5 (2.88)
  Day 1, 12 hour | 0.4 (2.37) | -0.5 (1.76) | 0.0 (3.22) | 0.8 (2.40) | 0.8 (1.72) | 0.5 (3.56)
  Day 1, 16 hour | -0.4 (2.22) | -1.8 (2.14) | -1.3 (2.25) | 0.0 (3.35) | 0.7 (1.75) | -0.8 (2.23)
  Day 2 | -0.3 (1.70) | 0.2 (1.60) | -0.3 (0.82) | -0.5 (2.95) | 1.5 (2.17) | -0.3 (3.01)
  Day 3 | 0.4 (1.90) | -0.3 (1.97) | 0.3 (3.56) | 0.3 (2.07) | 1.3 (2.34) | -0.2 (2.40)
  Day 4 | 0.6 (2.01) | -0.2 (1.72) | -0.5 (2.26) | -0.5 (2.51) | 0.5 (2.07) | -0.2 (2.56)
  Day 5 | 0.4 (0.97) | -0.7 (1.21) | 0.5 (3.27) | 1.5 (1.76) | 0.8 (1.47) | 0.3 (3.61)
  Day 7 | 0.3 (1.89) | -0.3 (1.21) | -0.5 (1.87) | 0.5 (2.07) | -0.3 (1.86) | 0.5 (2.07)

6. Primary Outcome: Number of Participants With Hematology Parameters Outside Reference Range Part 1
Description: Hematology parameters included hemoglobin (HGB), hematocrit (HCT), Red Blood Cell (RBC) count, White Blood Cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH) and mean corpuscular hemoglobin concentration (MCHC). Reference range for basophil was 0.01 - 0.07*10^9/Liters (L), eosinophils 0.03 - 0.5*10^9/L, HCT 0.38 - 0.48 proportion of RBC in blood, HGB 126 - 165*gram (g)/L, lymphocytes 1.08 - 3*10^9/L, MCH 26.3 - 32.8*picogram (pg), MCHC 324 - 359*g/L, MCV 77 - 94.9*femtoliter (fL), monocytes 0.3 - 0.92*10^9/L, neutrophils 1.46 - 5.85*10^9/L, platelets 155 - 342*10^9/L, erythrocytes 4.12 - 5.74*10^12/L, leukocytes 3.19 - 8.71*10^9/L. Values below these ranges were considered as low and above these ranges were considered as high (H). Data for participants from any visit post-screening with values > reference range high and < reference range low are report.
Time Frame: Up to Day 7
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Basophil, > reference range H | 0 | 0 | 0 | 0 | 0 | 1
  Basophil, < reference range low | 1 | 0 | 0 | 0 | 0 | 0
  Eosinophils, > reference range H | 0 | 0 | 2 | 0 | 0 | 1
  Eosinophils, < reference range low | 2 | 0 | 0 | 0 | 0 | 2
  MCHC, > reference range H | 1 | 0 | 0 | 0 | 0 | 0
  MCHC,< reference range low | 0 | 0 | 1 | 0 | 1 | 0
  MCH, > reference range H | 0 | 2 | 1 | 0 | 1 | 1
  MCH, < reference range low | 0 | 0 | 1 | 0 | 1 | 1
  MCV, > reference range H | 2 | 1 | 2 | 0 | 0 | 0
  MCV, < reference range low | 0 | 0 | 1 | 0 | 1 | 0
  Erythrocytes, > reference range H | 0 | 0 | 1 | 0 | 0 | 0
  Erythrocytes, < reference range low | 1 | 1 | 0 | 0 | 0 | 0
  HCT,> reference range H | 1 | 0 | 0 | 0 | 0 | 0
  HCT, < reference range low | 1 | 1 | 0 | 1 | 1 | 0
  HGB,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  HGB, < reference range low | 0 | 0 | 1 | 0 | 1 | 0
  Leukocytes,> reference range H | 1 | 1 | 5 | 4 | 5 | 5
  Leukocytes, < reference range low | 1 | 0 | 0 | 2 | 1 | 3
  Lymphocytes,> reference range H | 3 | 1 | 0 | 0 | 0 | 0
  Lymphocytes, < reference range low | 1 | 3 | 3 | 6 | 6 | 6
  Monocytes,> reference range H | 0 | 0 | 2 | 0 | 0 | 0
  Monocytes, < reference range low | 4 | 4 | 5 | 6 | 6 | 6
  Neutrophils,> reference range H | 0 | 0 | 5 | 4 | 5 | 6
  Neutrophils, < reference range low | 2 | 0 | 1 | 1 | 1 | 3
  Platelets,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, < reference range low | 1 | 3 | 0 | 0 | 1 | 1

7. Primary Outcome: Number of Participants With Clinical Chemistry Parameters Outside Reference Range
Description: Clinical chemistry parameters with reference range were albumin 35-52*g/L, Alkaline phosphatase (ALP) 30-120*International units/L (IU/L), Alanine aminotransferase (ALT) 0-50 * IU/L, Aspartate aminotransferase (AST) 0-50*IU/L, direct bilirubin 0-3.4* micromoles/L (µmol/L), bilirubin 5-21*µmol/L, calcium 2.2-2.65* millimoles/L (mmol/L), cholesterol 0-5.19* mmol/L, creatinine 59-104* µmol/L, C-reactive protein (CRP) 0-5*milligram (mg)/L,Gamma Glutamyl Transferase (GGT) 4.1-5.9*mmol/L, high density lipoproteins (HDL) cholesterol 0.99-2.32*mmol/L, potassium 3.5-5.1*mmol/L, low density lipoproteins (LDL) cholesterol 0-3.3*mmol/L, protein 66-83*g/L, sodium 136-146 * mmol/L, triglycerides 0-2.25 * mmol/L, glucose 4.1-5.9*mmol/L, and urea 2.8-7.2*mmol/L. Values below these ranges were considered as low and above these ranges were considered as high. Data for participants from any visit post-screening with values > reference range high and < reference range low are reported.
Time Frame: Up to Day 7
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  ALT, > reference range H | 0 | 0 | 2 | 0 | 1 | 0
  ALT, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, > reference range H | 00 | 0 | 0 | 0 | 0 | 0
  Albumin, < reference range low | 0 | 0 | 0 | 1 | 0 | 0
  ALP, > reference range H | 0 | 0 | 0 | 0 | 0 | 0
  ALP,< reference range low | 0 | 0 | 0 | 0 | 0 | 0
  AST, > reference range H | 0 | 0 | 0 | 1 | 0 | 0
  AST, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, > reference range H | 2 | 1 | 0 | 0 | 0 | 0
  Bilirubin, < reference range low | 3 | 0 | 0 | 1 | 0 | 0
  CRP, > reference range H | 1 | 0 | 2 | 4 | 5 | 6
  CRP, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Calcium,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, < reference range low | 1 | 0 | 1 | 1 | 2 | 2
  Creatinine,> reference range H | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine, < reference range low | 1 | 0 | 1 | 0 | 0 | 1
  Direct Bilirubin,> reference range H | 1 | 1 | 0 | 0 | 0 | 0
  Direct Bilirubin, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Glucose,> reference range H | 0 | 0 | 2 | 0 | 0 | 0
  Glucose, < reference range low | 0 | 0 | 0 | 2 | 0 | 1
  Indirect bilirubin,> reference range H | 1 | 0 | 0 | 0 | 0 | 0
  Indirect bilirubin, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Potassium,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, < reference range low | 0 | 0 | 0 | 0 | 0 | 0
  Protein,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  Protein, < reference range low | 4 | 4 | 3 | 4 | 4 | 5
  Sodium,> reference range H | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, < reference range low | 2 | 2 | 3 | 2 | 3 | 3
  Urea,> reference range H | 0 | 1 | 0 | 0 | 0 | 0
  Urea, < reference range low | 1 | 1 | 1 | 1 | 1 | 0

8. Primary Outcome: Casts, Round Epithelial Cells (REC), Squamous Epithelial Cells (SEC), Urine Erythrocytes and Urine Leukocytes at Indicated Time Points
Description: Urinalysis included microscopic examination parameters like Casts, REC, SEC, Urine erythrocytes and Urine leukocytes. Data at indicated time points were reported. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles). NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point.
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Cells per high power field
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Cells per high power field
  Casts, Day -1 Pre-dose, n=1,0,2,1,0,1: number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 1
  Casts, Day -1 Pre-dose, n=1,0,2,1,0,1 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. |  | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. |  | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point.
  Casts, Day 1, Pre-dose, n=3,1,2,0,0,2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0 | 2
  Casts, Day 1, Pre-dose, n=3,1,2,0,0,2 | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. | 0.0 (0.0) |  |  | 0.0 (0.0)
  Casts, Day 2, n=1,0,3,1,1,2: number analyzed (Participants) | 1 | 0 | 3 | 1 | 1 | 2
  Casts, Day 2, n=1,0,3,1,1,2 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. |  | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. | 0.0 (0.0)
  Casts, Day 4, n=3,0,1,2,0,0: number analyzed (Participants) | 3 | 0 | 1 | 2 | 0 | 0
  Casts, Day 4, n=3,0,1,2,0,0 | 0.0 (0.0) |  | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point. | 0.0 (0.0) |  |
  Casts, Day 7, n=4,0,2,2,0,0: number analyzed (Participants) | 4 | 0 | 2 | 2 | 0 | 0
  Casts, Day 7, n=4,0,2,2,0,0 | 0.0 (0.0) |  | 0.0 (0.0) | 0.0 (0.0) |  |
  REC, Day -1 Pre-dose, n=1,0,2,1,0,1: number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 1
  REC, Day -1 Pre-dose, n=1,0,2,1,0,1 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point
  REC, Day 1 Pre-dose, n=3,1,2,0,0,2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0 | 2
  REC, Day 1 Pre-dose, n=3,1,2,0,0,2 | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0) |  |  | 0.0 (0.0)
  REC, Day 2 , n=1,0,3,1,1,2: number analyzed (Participants) | 1 | 0 | 3 | 1 | 1 | 2
  REC, Day 2 , n=1,0,3,1,1,2 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0)
  REC, Day 4, n=3,0,1,2,0,0: number analyzed (Participants) | 3 | 0 | 1 | 2 | 0 | 0
  REC, Day 4, n=3,0,1,2,0,0 | 0.0 (0.0) |  | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0) |  |
  REC, Day 7, n=4,0,2,2,0,0: number analyzed (Participants) | 4 | 0 | 2 | 2 | 0 | 0
  REC, Day 7, n=4,0,2,2,0,0 | 0.0 (0.0) |  | 0.0 (0.0) | 0.0 (0.0) |  |
  SEC, Day -1 Pre-dose, n=1,0,2,1,0,1: number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 1
  SEC, Day -1 Pre-dose, n=1,0,2,1,0,1 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 4.0 (5.66) | 8.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 3.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point
  SEC, Day 1 Pre-dose, n=3,1,2,0,0,2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0 | 2
  SEC, Day 1 Pre-dose, n=3,1,2,0,0,2 | 1.0 (1.73) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 2.0 (2.83) |  |  | 1.5 (0.71)
  SEC, Day 2 , n=1,0,3,1,1,2: number analyzed (Participants) | 1 | 0 | 3 | 1 | 1 | 2
  SEC, Day 2 , n=1,0,3,1,1,2 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (0.0) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0)
  SEC, Day 4, n=3,0,1,2,0,0: number analyzed (Participants) | 3 | 0 | 1 | 2 | 0 | 0
  SEC, Day 4, n=3,0,1,2,0,0 | 0.0 (0.0) |  | 10.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 1.0 (1.41) |  |
  SEC, Day 7, n=4,0,2,2,0,0: number analyzed (Participants) | 4 | 0 | 2 | 2 | 0 | 0
  SEC, Day 7, n=4,0,2,2,0,0 | 1.5 (3.00) |  | 0.0 (0.0) | 11.0 (12.73) |  |
  Urine Erythrocytes,Day -1 Pre-dose, n=1,0,2,1,0,1: number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 1
  Urine Erythrocytes,Day -1 Pre-dose, n=1,0,2,1,0,1 | 5.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.5 (0.71) | 3.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 1.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point
  Urine Erythrocytes,Day 1 Pre-dose, n=3,1,2,0,0,2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0 | 2
  Urine Erythrocytes,Day 1 Pre-dose, n=3,1,2,0,0,2 | 2.3 (4.04) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0) |  |  | 0.0 (0.0)
  Urine Erythrocytes,Day 2 , n=1,0,3,1,1,2: number analyzed (Participants) | 1 | 0 | 3 | 1 | 1 | 2
  Urine Erythrocytes,Day 2 , n=1,0,3,1,1,2 | 1.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (0.0) | 7.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.5 (0.71)
  Urine Erythrocytes,Day 4, n=3,0,1,2,0,0: number analyzed (Participants) | 3 | 0 | 1 | 2 | 0 | 0
  Urine Erythrocytes,Day 4, n=3,0,1,2,0,0 | 1.0 (1.00) |  | 2.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (0.0) |  |
  Urine Erythrocytes,Day 7, n=4,0,2,2,0,0: number analyzed (Participants) | 4 | 0 | 2 | 2 | 0 | 0
  Urine Erythrocytes,Day 7, n=4,0,2,2,0,0 | 0.5 (1.00) |  | 0.0 (0.0) | 0.0 (0.0) |  |
  Urine Leukocytes,Day -1 Pre-dose, n=1,0,2,1,0,1: number analyzed (Participants) | 1 | 0 | 2 | 1 | 0 | 1
  Urine Leukocytes,Day -1 Pre-dose, n=1,0,2,1,0,1 | 1.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 1.5 (2.12) | 1.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 4.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point
  Urine Leukocytes,Day 1 Pre-dose, n=3,1,2,0,0,2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 0 | 2
  Urine Leukocytes,Day 1 Pre-dose, n=3,1,2,0,0,2 | 5.0 (8.66) | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.5 (0.71) |  |  | 3.0 (2.83)
  Urine Leukocytes,Day 2 , n=1,0,3,1,1,2: number analyzed (Participants) | 1 | 0 | 3 | 1 | 1 | 2
  Urine Leukocytes,Day 2 , n=1,0,3,1,1,2 | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point |  | 0.0 (0.0) | 4.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 0.5 (0.71)
  Urine Leukocytes,Day 4, n=3,0,1,2,0,0: number analyzed (Participants) | 3 | 0 | 1 | 2 | 0 | 0
  Urine Leukocytes,Day 4, n=3,0,1,2,0,0 | 1.0 (1.73) |  | 3.0 (NA) — NA indicates standard deviation could not be calculated as only 1 participant was analyzed at the given time point | 42.0 (59.40) |  |
  Urine Leukocytes,Day 7, n=4,0,2,2,0,0: number analyzed (Participants) | 4 | 0 | 2 | 2 | 0 | 0
  Urine Leukocytes,Day 7, n=4,0,2,2,0,0 | 0.3 (0.50) |  | 0.0 (0.0) | 40.5 (55.86) |  |

9. Primary Outcome: Ketones and Urine Glucose at Indicated Time Points
Description: Urinalysis included parameters like ketones and urine glucose. Data at indicated time points were reported.
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Millimoles per liter
  Ketones, Pre-dose Day -1 | 0.05 (0.158) | 0.00 (0.000) | 0.08 (0.204) | 0.00 (0.000) | 0.00 (0.000) | 0.25 (0.612)
  Ketones, Pre-dose Day 1 | 0.05 (0.158) | 0.00 (0.000) | 0.25 (0.612) | 0.00 (0.000) | 0.00 (0.000) | 0.08 (0.204)
  Ketones, Day 2 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.00) | 0.00 (0.000) | 0.00 (0.000) | 1.75 (2.525)
  Ketones, Day 4 | 0.15 (0.242) | 0.00 (0.000) | 0.08 (0.204) | 0.00 (0.000) | 0.00 (0.000) | 0.08 (0.204)
  Ketones, Day 7 | 0.00 (0.000) | 0.00 (0.000) | 0.08 (0.204) | 0.25 (0.612) | 0.00 (0.000) | 0.08 (0.204)
  Urine glucose, Pre-dose Day -1 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Urine glucose, Pre-dose Day 1 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Urine glucose, Day 2 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Urine glucose, Day 4 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Urine glucose, Day 7 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

10. Primary Outcome: Occult Blood at Indicated Time Points
Description: Urinalysis included parameter like Occult blood. Data at indicated time points were reported.
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
10^9 cells per liter
  Pre-dose Day -1 | 2.5 (7.91) | 0.0 (0.00) | 5.8 (10.21) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Pre-dose Day 1 | 4.5 (8.32) | 1.7 (4.08) | 3.3 (5.16) | 0.0 (0.00) | 0.0 (0.00) | 1.7 (4.08)
  Day 2 | 2.5 (7.91) | 0.0 (0.00) | 5.0 (5.48) | 4.2 (10.21) | 1.7 (4.08) | 5.8 (10.21)
  Day 4 | 4.5 (8.32) | 0.0 (0.00) | 0.0 (0.00) | 4.2 (10.21) | 0.0 (0.00) | 0.0 (0.00)
  Day 7 | 4.0 (5.16) | 0.0 (0.00) | 8.3 (12.91) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

11. Primary Outcome: Urine Protein at Indicated Time Points
Description: Urinalysis included parameter like Urine protein. Data at indicated time points were reported.
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Gram per liter
  Pre-dose Day -1 | 0.000 (0.0000) | 0.000 (0.0000) | 0.042 (0.1021) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Pre-dose Day 1 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 2 | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 4 | 0.025 (0.0791) | 0.000 (0.0000) | 0.042 (0.1021) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 7 | 0.000 (0.0000) | 0.000 (0.0000) | 0.042 (0.1021) | 0.042 (0.1021) | 0.000 (0.0000) | 0.000 (0.0000)

12. Primary Outcome: Specific Gravity at Indicated Time Points
Description: Urinalysis included parameter like specific gravity. Urinary specific gravity is a measure of the concentration of solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine.
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Ratio
  Pre-dose Day -1 | 1.018 (0.0065) | 1.008 (0.0053) | 1.017 (0.0091) | 1.015 (0.0019) | 1.008 (0.0030) | 1.019 (0.0047)
  Pre-dose Day 1 | 1.014 (0.0072) | 1.011 (0.0048) | 1.015 (0.0083) | 1.013 (0.0063) | 1.008 (0.0031) | 1.014 (0.0060)
  Day 2 | 1.017 (0.0049) | 1.013 (0.0055) | 1.017 (0.0041) | 1.016 (0.0044) | 1.014 (0.0048) | 1.017 (0.0072)
  Day 4 | 1.019 (0.0069) | 1.014 (0.0041) | 1.018 (0.0072) | 1.016 (0.0038) | 1.014 (0.0061) | 1.016 (0.0059)
  Day 7 | 1.016 (0.0082) | 1.006 (0.0025) | 1.015 (0.0117) | 1.015 (0.0090) | 1.010 (0.0079) | 1.013 (0.0058)

13. Primary Outcome: Urine Potential of Hydrogen (pH) at Indicated Time Points
Description: Urinalysis parameters included urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0).
Time Frame: Pre-dose Day -1 and Day 1, Day 2, Day 4 and Day 7
Population: All Subject Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
pH
  Pre-dose Day -1 | 6.10 (0.843) | 6.42 (0.801) | 5.00 (0.000) | 5.83 (0.931) | 6.50 (0.775) | 5.67 (0.753)
  Pre-dose Day 1 | 6.05 (0.926) | 5.83 (0.931) | 5.75 (0.822) | 5.50 (0.837) | 6.25 (0.758) | 5.33 (0.816)
  Day 2 | 6.20 (0.753) | 5.83 (0.983) | 5.92 (0.801) | 6.25 (0.689) | 5.33 (0.516) | 5.50 (0.837)
  Day 4 | 5.95 (0.725) | 5.67 (1.033) | 5.50 (0.775) | 5.92 (1.021) | 6.08 (0.917) | 5.67 (0.816)
  Day 7 | 6.00 (0.882) | 5.58 (0.917) | 5.25 (0.612) | 5.75 (0.880) | 5.92 (0.801) | 6.08 (0.917)

14. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECG) Findings Worst Case Post-Baseline
Description: Single measurements of 12-lead ECGs were obtained after 10 minutes of rest in a semi-supine position for the participant. Participants with abnormal ECG findings that are clinically not significant (NCS) and clinically significant (CS) data has been presented here. The data of worst case post-Baseline is presented here.
Time Frame: Up to Day 32
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  NCS | 3 | 1 | 1 | 2 | 1 | 1
  CS | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of GSK1795091 for Part 1
Description: Blood samples were collected at indicated time points. The Pharmacokinetic (PK) parameters were calculated for each participant using a non-compartmental method. All participants for whom, at least, one valid and evaluable pharmacokinetic parameter (AUC or Cmax) was derived were included in PK Parameter Population. Only those participants with data available at the specified data points were analyzed.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: PK Parameter Population. NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram/milliliter (pg/mL)
Arm/Group | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Picogram/milliliter (pg/mL) | NA (NA) — NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification. | 3.78 (15.9) | 10.1 (13.0) | 9.45 (25.5) | 23.7 (6.69)

16. Secondary Outcome: Time of Occurrence of Cmax (Tmax) and Terminal Half Life (t1/2) of GSK1795091 for Part 1
Description: Blood samples were collected at indicated time points. The PK parameters were calculated for each participant using a non-compartmental method. Only those participants with data available at the specified data points were analyzed.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Hours
  t1/2 | NA (NA) — NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification. | 25.2 (9.51) | 45.7 (12.5) | 67.1 (33.9) | 69.4 (9.24)
  tmax | NA (NA) — NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification. | 0.0950 (0.0197) | 0.0833 (0.00816) | 0.103 (0.0755) | 0.0880 (0.0110)

17. Secondary Outcome: Partial Area Under the Concentration-time Curve to Time t (AUC[0-t]), Area Under the Concentration-time Curve (AUC) From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of GSK1795091 for Part 1
Description: Blood samples were collected at indicated time points. The PK parameters were calculated for each participant using a non-compartmental method. AUC (0-t) was used interchangeably with AUC to last time of quantifiable concentration (AUC[0-last]) .Only those participants with data available at the specified data points were analyzed.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: PK Parameter Population. NA indicates data was not available as all concentration outcomes at 7ng were not quantifiable because all results were below the limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*pg/mL
Arm/Group | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Hours*pg/mL
  AUC(0-t) | NA (NA) — NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification. | 21.1 (89.7) | 233 (56.4) | 264 (33.3) | 1100 (12.2)
  AUC(0-inf) | NA (NA) — NA indicates data was not available for 7 ng Arm as all concentration outcomes at 7 ng were not quantifiable because all results were below the limit of quantification. | 104 (52.2) | 417 (40.0) | 532 (26.3) | 1440 (15.9)

18. Secondary Outcome: Clearance (CL) of GSK1795091 for Part 1
Description: as for outcome 16
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Liters per hour (L/h) | NA (NA) — NA indicates data was not available as all concentration outcomes at 7ng were not quantifiable because all results were below the limit of quantification. | 0.202 (52.2) | 0.144 (40.0) | 0.113 (26.3) | 0.0693 (15.9)

19. Secondary Outcome: Volume of Distribution of GSK1795091 for Part 1
Description: as for outcome 16
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Liters (L) | NA (NA) — NA indicates data was not available as all concentration outcomes at 7ng were not quantifiable because all results were below the limit of quantification. | 6.95 (10.1) | 9.46 (24.2) | 9.95 (25.7) | 6.75 (10.7)

20. Secondary Outcome: Percentage Fold Change of Concentration of Interleukin 6 (IL-6) From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of IL-6. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline. All participants in the "All Subjects Population" for whom valid and evaluable pharmacodynamic parameters were derived are included in Pharmacodynamic (PD) Population. Data from multiplex immunoassay has been reported.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population.
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | 40.17 (51.192) | 30.81 (33.517) | 193.49 (163.904) | 332.92 (310.845) | 588.11 (324.942) | 956.69 (763.404)
  2 hour | 26.49 (39.212) | 239.27 (301.767) | 625.51 (547.296) | 1801.82 (1788.852) | 2171.25 (1363.074) | 7305.11 (6138.721)
  4 hour | 169.63 (421.394) | 255.33 (254.874) | 513.81 (523.303) | 803.37 (1020.453) | 1244.12 (1759.562) | 1170.88 (767.439)
  8 hour | 262.38 (339.956) | 161.33 (187.908) | 338.13 (317.030) | 166.86 (176.423) | 677.24 (903.777) | 190.07 (181.963)
  12 hour | 267.01 (274.112) | 832.13 (965.345) | 938.35 (1585.370) | 500.75 (827.894) | 644.77 (311.661) | 363.91 (610.090)
  16 hour | 284.52 (356.147) | 607.83 (986.760) | 249.04 (280.046) | 467.74 (620.968) | 326.81 (300.766) | 210.55 (425.106)
  24 hour | 129.34 (110.041) | 200.07 (261.810) | 56.24 (157.132) | 182.47 (248.911) | 201.93 (375.976) | 160.58 (383.092)
  48 hour | -13.13 (46.097) | -33.21 (30.172) | -18.95 (45.030) | -21.89 (30.042) | -14.22 (42.014) | -26.67 (21.931)
  144 hour | -12.48 (27.665) | -29.63 (38.535) | -19.58 (26.650) | -4.52 (41.111) | -10.87 (26.937) | -6.59 (39.036)

21. Secondary Outcome: Percentage Fold Change of Concentration of Tumor Necrosis Factor (TNF)-Alpha From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of TNF-alpha. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline. Data from multiplex immunoassay has been reported. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population.
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  1 hour, n=8, 3, 5, 5, 4, 5 | 3.61 (28.753) | 12.51 (22.453) | 112.63 (185.111) | 130.88 (126.286) | 771.06 (579.613) | 1838.09 (2790.783)
  2 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  2 hour, n=8, 3, 5, 5, 4, 5 | -1.26 (11.879) | -6.42 (5.229) | 209.17 (437.355) | 51.85 (58.482) | 379.87 (299.578) | 661.61 (998.133)
  4 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  4 hour, n=8, 3, 5, 5, 4, 5 | -4.38 (12.448) | -5.82 (8.277) | 164.74 (402.327) | 12.90 (22.215) | 66.55 (76.017) | 18.87 (26.716)
  8 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  8 hour, n=8, 3, 5, 5, 4, 5 | 1.72 (8.690) | -12.56 (13.872) | 75.34 (202.570) | 2.28 (4.332) | 11.12 (32.576) | -7.87 (10.985)
  12 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  12 hour, n=8, 3, 5, 5, 4, 5 | 4.38 (19.376) | -10.33 (26.632) | 54.30 (170.246) | 7.61 (10.968) | 24.14 (35.746) | -4.21 (9.459)
  16 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  16 hour, n=8, 3, 5, 5, 4, 5 | -1.81 (17.321) | -11.77 (16.419) | 17.36 (92.732) | -1.28 (9.826) | 43.11 (90.323) | -11.41 (14.569)
  24 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  24 hour, n=8, 3, 5, 5, 4, 5 | 3.30 (30.223) | -10.02 (21.221) | 17.39 (75.367) | 7.26 (13.568) | 34.79 (37.921) | -6.04 (17.245)
  48 hour, n=8, 3, 5, 5, 3, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 3 | 5
  48 hour, n=8, 3, 5, 5, 3, 5 | -2.56 (16.028) | -7.18 (9.567) | -10.99 (37.153) | 4.03 (23.030) | -2.31 (45.586) | -13.33 (14.853)
  144 hour, n=8, 3, 5, 5, 4, 5: number analyzed (Participants) | 8 | 3 | 5 | 5 | 4 | 5
  144 hour, n=8, 3, 5, 5, 4, 5 | -7.34 (15.006) | -2.90 (20.283) | -14.85 (27.169) | -2.10 (37.702) | 5.46 (31.910) | -5.16 (17.479)

22. Secondary Outcome: Percentage Fold Change of Concentration of Interferon (IFN)-Gamma From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of IFN-gamma. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline. Data from multiplex immunoassay has been reported. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour, n=9, 5, 4, 6, 6, 5: number analyzed (Participants) | 9 | 5 | 4 | 6 | 6 | 5
  1 hour, n=9, 5, 4, 6, 6, 5 | -1.24 (7.942) | -6.31 (7.547) | -3.16 (6.918) | -1.52 (3.299) | -8.15 (9.430) | 14.42 (17.175)
  2 hour, n=10, 5, 4, 6, 6, 5: number analyzed (Participants) | 10 | 5 | 4 | 6 | 6 | 5
  2 hour, n=10, 5, 4, 6, 6, 5 | 5.04 (13.885) | -7.35 (10.068) | -0.81 (4.453) | 17.81 (56.864) | 72.02 (125.017) | 104.54 (208.806)
  4 hour, n=10, 5, 4, 6, 6, 5: number analyzed (Participants) | 10 | 5 | 4 | 6 | 6 | 5
  4 hour, n=10, 5, 4, 6, 6, 5 | -2.39 (8.391) | 2.33 (6.932) | 49.66 (97.641) | 119.86 (211.426) | 247.58 (188.954) | 229.73 (352.909)
  8 hour, n=10, 5, 4, 6, 6, 5: number analyzed (Participants) | 10 | 5 | 4 | 6 | 6 | 5
  8 hour, n=10, 5, 4, 6, 6, 5 | 0.05 (5.453) | -0.10 (5.957) | 13.68 (39.549) | 36.75 (48.057) | 86.13 (63.258) | 66.69 (94.960)
  12 hour, n=10, 5, 4, 6, 6, 5: number analyzed (Participants) | 10 | 5 | 4 | 6 | 6 | 5
  12 hour, n=10, 5, 4, 6, 6, 5 | 4.48 (14.140) | -7.01 (27.233) | -9.18 (10.540) | 20.90 (32.530) | 38.35 (48.687) | 31.00 (37.179)
  16 hour, n=10, 5, 4, 6, 6, 5: number analyzed (Participants) | 10 | 5 | 4 | 6 | 6 | 5
  16 hour, n=10, 5, 4, 6, 6, 5 | 6.51 (24.803) | -6.27 (29.923) | -15.42 (22.050) | 20.62 (29.976) | 34.82 (46.979) | 12.75 (19.418)
  24 hour, n=10, 4, 4, 6, 6, 5: number analyzed (Participants) | 10 | 4 | 4 | 6 | 6 | 5
  24 hour, n=10, 4, 4, 6, 6, 5 | 3.96 (17.217) | 6.57 (16.853) | -19.32 (32.943) | 2.48 (8.071) | -3.08 (14.045) | 6.46 (8.403)
  48 hour, n=10, 4, 4, 6, 6, 5: number analyzed (Participants) | 10 | 4 | 4 | 6 | 6 | 5
  48 hour, n=10, 4, 4, 6, 6, 5 | 4.21 (22.768) | 1.41 (6.871) | -19.82 (34.669) | -3.63 (13.448) | 0.39 (20.837) | 2.43 (5.216)
  144 hour, n=10, 4, 3, 6, 6, 5: number analyzed (Participants) | 10 | 4 | 3 | 6 | 6 | 5
  144 hour, n=10, 4, 3, 6, 6, 5 | 33.01 (107.893) | 4.96 (8.947) | -2.15 (13.149) | -4.16 (14.851) | 6.81 (21.544) | -1.26 (5.652)

23. Secondary Outcome: Percentage Fold Change of Concentration of Inducible Protein (IP)-10 From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of IP-10. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | -17.09 (11.676) | -22.96 (9.621) | -10.99 (11.237) | -21.97 (10.771) | -6.50 (12.551) | 14.49 (35.063)
  2 hour | -15.30 (9.675) | -8.75 (16.126) | 39.93 (26.514) | 54.49 (58.967) | 112.79 (66.958) | 312.12 (121.798)
  4 hour | -14.34 (11.025) | 25.43 (42.934) | 351.07 (286.393) | 1672.77 (1676.676) | 2045.12 (1937.378) | 6740.10 (1888.455)
  8 hour | -11.97 (10.564) | 4.07 (29.521) | 119.48 (103.465) | 338.47 (349.007) | 538.99 (614.669) | 2367.11 (1067.103)
  12 hour | -22.97 (8.906) | -9.76 (17.265) | 46.78 (40.980) | 133.47 (128.186) | 337.37 (416.181) | 802.21 (272.436)
  16 hour | -14.51 (14.185) | -6.75 (20.215) | 52.55 (32.122) | 99.47 (114.305) | 238.17 (321.382) | 394.46 (171.075)
  24 hour | -2.89 (20.587) | 25.65 (38.100) | 46.42 (25.692) | 67.34 (34.573) | 137.55 (128.045) | 186.87 (57.860)
  48 hour | 6.24 (28.068) | 37.30 (78.673) | 31.98 (40.635) | 35.61 (26.802) | 41.03 (42.609) | 57.44 (28.805)
  144 hour | 5.97 (35.519) | 20.56 (41.682) | 16.66 (39.635) | 15.62 (50.973) | 24.18 (21.117) | 29.64 (21.330)

24. Secondary Outcome: Percentage Fold Change of Concentration of Monocyte Chemotactic Protein 1 (MCP-1) From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of MCP-1. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | 0.39 (9.459) | -1.15 (10.591) | 4.50 (12.165) | 18.59 (24.366) | 21.31 (30.421) | 119.24 (58.836)
  2 hour | 0.73 (9.124) | 76.83 (60.093) | 481.09 (255.487) | 1097.31 (743.475) | 2604.72 (1691.082) | 5883.27 (2461.263)
  4 hour | -3.44 (14.828) | 64.60 (54.045) | 315.88 (237.902) | 907.01 (928.980) | 1241.68 (1744.836) | 5290.85 (2834.623)
  8 hour | 1.97 (14.914) | 7.94 (17.127) | 35.25 (25.294) | 51.16 (29.055) | 70.82 (58.048) | 223.95 (113.142)
  12 hour | 6.99 (16.748) | 16.17 (18.245) | 29.60 (25.748) | 32.76 (23.618) | 56.45 (56.466) | 111.19 (67.497)
  16 hour | 11.29 (17.046) | 29.40 (25.521) | 26.43 (9.956) | 35.30 (25.461) | 39.71 (40.794) | 45.49 (18.571)
  24 hour | -6.26 (9.139) | -1.42 (9.045) | 4.06 (7.179) | -7.95 (11.240) | 3.90 (14.549) | 10.69 (16.458)
  48 hour | -3.16 (12.267) | -1.40 (9.991) | -1.51 (9.848) | -8.02 (15.104) | -7.40 (10.834) | -3.58 (10.363)
  144 hour | 13.23 (20.203) | 24.53 (11.806) | 22.01 (11.379) | 8.74 (24.846) | 14.97 (16.939) | 15.23 (12.460)

25. Secondary Outcome: Percentage Fold Change of Colony Stimulating Factor 2 (GCSF) From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of GCSF. Baseline was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | -0.99 (5.692) | -4.68 (10.515) | 2.58 (7.662) | 2.91 (16.607) | 5.83 (8.244) | 25.99 (11.220)
  2 hour | 2.91 (6.204) | 2.69 (12.149) | 11.12 (11.405) | 162.85 (247.315) | 105.64 (96.885) | 1365.60 (893.674)
  4 hour | 10.78 (18.117) | 4.38 (9.022) | 13.23 (15.291) | 933.31 (1826.357) | 390.62 (541.504) | 3754.71 (2439.913)
  8 hour | 19.67 (23.987) | 16.22 (12.747) | 9.78 (24.467) | 150.61 (232.289) | 96.07 (123.200) | 595.98 (316.686)
  12 hour | 16.42 (20.532) | 13.85 (17.900) | 8.85 (20.773) | 71.44 (71.786) | 59.51 (72.401) | 265.40 (166.832)
  16 hour | 5.83 (13.164) | 10.84 (18.000) | -2.49 (17.532) | 30.82 (39.981) | 22.29 (55.206) | 162.78 (121.912)
  24 hour | 6.67 (9.270) | 4.50 (13.016) | 1.23 (10.457) | 23.82 (29.497) | 15.76 (36.063) | 96.88 (87.031)
  48 hour | 6.29 (12.038) | 2.52 (10.170) | -1.26 (10.068) | 19.14 (17.687) | 3.08 (25.153) | 17.08 (32.119)
  144 hour | 4.74 (19.231) | -10.01 (13.393) | 7.06 (23.343) | -4.23 (16.821) | -5.25 (21.081) | -4.94 (23.010)

26. Secondary Outcome: Percentage Fold Change of Interleukin 1 Receptor Antagonist (IL-1Ra) From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of IL-1Ra. Baseline was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | 4.06 (12.046) | -1.63 (15.193) | 11.49 (8.978) | 19.88 (23.137) | 38.00 (20.565) | 111.99 (25.295)
  2 hour | 5.26 (17.249) | 26.95 (19.100) | 149.20 (53.633) | 607.17 (611.511) | 803.47 (486.468) | 7054.40 (1029.027)
  4 hour | 13.43 (24.391) | 196.62 (186.603) | 1716.81 (1046.690) | 12062.23 (13307.136) | 13359.29 (9271.512) | 105032.57 (61423.988)
  8 hour | 20.78 (28.762) | 103.59 (63.317) | 818.24 (578.438) | 3136.61 (3429.187) | 2788.30 (2101.015) | 16830.47 (7106.072)
  12 hour | 21.64 (23.580) | 99.49 (75.059) | 360.87 (233.664) | 1207.18 (1324.133) | 1422.66 (1254.465) | 7055.35 (3496.863)
  16 hour | 29.17 (28.404) | 61.72 (38.867) | 217.81 (154.263) | 524.89 (652.117) | 723.30 (718.195) | 2273.75 (783.885)
  24 hour | 35.02 (51.217) | 19.31 (36.307) | 75.80 (64.742) | 124.90 (154.983) | 195.35 (136.345) | 400.73 (98.553)
  48 hour | -11.07 (23.224) | -3.86 (13.848) | 10.45 (25.851) | 7.64 (28.049) | 15.71 (18.469) | 37.51 (17.058)
  144 hour | -2.00 (35.912) | -0.95 (19.617) | -2.03 (19.870) | 3.17 (33.828) | 3.26 (14.855) | 2.75 (13.556)

27. Secondary Outcome: Percentage Fold Change of Interleukin 10 (IL-10) From Baseline for Part 1
Description: Blood samples were collected at indicated time points for the assessment of IL-10. Baseline was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Percentage fold change equals to 100*change from Baseline divided by Baseline.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population
Measure: Mean (Standard Deviation); unit: Percent fold change
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 5
Percent fold change
  1 hour | 4.18 (2.923) | 36.13 (50.565) | 131.03 (167.082) | 170.79 (130.626) | 320.02 (171.738) | 590.82 (378.761)
  2 hour | 3.89 (5.943) | 138.05 (233.654) | 496.20 (746.150) | 437.92 (436.690) | 587.14 (327.563) | 2985.38 (2768.658)
  4 hour | 7.66 (9.351) | 35.74 (39.419) | 72.32 (81.429) | 75.74 (75.003) | 104.81 (83.542) | 166.23 (149.184)
  8 hour | 1.45 (9.681) | 13.56 (22.309) | 44.31 (54.738) | 38.31 (30.005) | 98.31 (80.140) | 152.84 (125.207)
  12 hour | -0.94 (11.658) | 4.52 (18.393) | 22.10 (30.976) | 18.10 (20.319) | 39.32 (35.208) | 46.01 (29.984)
  16 hour | 8.81 (23.057) | 13.70 (20.597) | 23.52 (32.664) | 25.13 (19.212) | 48.07 (34.705) | 36.84 (22.787)
  24 hour | 14.43 (24.246) | 6.07 (9.298) | 11.37 (17.257) | 16.47 (10.573) | 24.70 (25.961) | 21.83 (17.997)
  48 hour | 13.20 (45.366) | 4.98 (5.925) | -1.41 (11.832) | 9.63 (5.995) | -0.10 (8.984) | 2.73 (10.103)
  144 hour | 17.99 (38.910) | 15.53 (13.540) | 10.35 (12.876) | 11.73 (4.742) | 14.73 (19.170) | 7.28 (10.035)

28. Secondary Outcome: Change From Baseline in WBC Differential for Part 1
Description: WBC differential included Lymphocytes Count, Monocytes Count, Granulocytes Count including neutrophils and eosinophil. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Time Frame: Baseline, 4, 24 and 144 hours
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
10^9 cells per liter
  Monocytes count, 4 hour, n=10, 6, 6, 5, 6, 6: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  Monocytes count, 4 hour, n=10, 6, 6, 5, 6, 6 | 0.012 (0.0543) | 0.156 (0.1228) | 0.253 (0.0759) | 0.129 (0.2242) | 0.169 (0.1512) | -0.061 (0.1629)
  Monocytes count, 24 hour, n=10, 6, 6, 6, 4, 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 4 | 6
  Monocytes count, 24 hour, n=10, 6, 6, 6, 4, 6 | 0.072 (0.1631) | -0.038 (0.1411) | 0.018 (0.0807) | 0.035 (0.1415) | 0.004 (0.0800) | 0.104 (0.3037)
  Monocytes count, 144 hour, n=10, 6, 6, 6, 6, 6 | 0.002 (0.0959) | 0.013 (0.1454) | -0.054 (0.0746) | 0.040 (0.1065) | -0.012 (0.0861) | -0.038 (0.0321)
  Granulocytes Count, 4 hour, n=10, 6, 6, 5, 6, 6: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  Granulocytes Count, 4 hour, n=10, 6, 6, 5, 6, 6 | 0.076 (0.2703) | 1.548 (0.8217) | 3.708 (0.8286) | 3.747 (2.3033) | 3.856 (0.8005) | 4.018 (4.9360)
  Granulocytes Count, 24 hour, n=10, 6, 6, 6, 4, 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 4 | 6
  Granulocytes Count, 24 hour, n=10, 6, 6, 6, 4, 6 | 0.400 (0.5482) | 0.062 (0.7474) | -0.691 (0.8687) | -0.122 (0.6265) | -0.176 (0.3004) | -0.940 (2.3939)
  Granulocytes Count, 144 hour, n=10, 6, 6, 6, 6, 6 | -0.067 (0.9350) | 0.292 (0.6764) | -0.669 (1.1381) | 0.245 (0.9796) | -0.073 (1.0629) | -0.974 (1.9877)
  Lymphocytes count, 4 hour, n=10, 6, 6, 5, 6, 6: number analyzed (Participants) | 10 | 6 | 6 | 5 | 6 | 6
  Lymphocytes count, 4 hour, n=10, 6, 6, 5, 6, 6 | 0.082 (0.2017) | -0.118 (0.3070) | -0.603 (0.2988) | -0.393 (0.7111) | -0.997 (0.4404) | -1.419 (1.3685)
  Lymphocytes count, 24 hour, n=10, 6, 6, 6, 4, 6: number analyzed (Participants) | 10 | 6 | 6 | 6 | 4 | 6
  Lymphocytes count, 24 hour, n=10, 6, 6, 6, 4, 6 | 0.135 (0.2034) | -0.045 (0.2957) | -0.051 (0.2327) | 0.042 (0.5468) | -0.247 (0.2634) | -0.489 (0.7405)
  Lymphocytes count, 144 hour, n=10, 6, 6, 6, 6, 6 | -0.080 (0.3950) | -0.107 (0.1786) | -0.030 (0.2490) | 0.060 (0.6556) | -0.175 (0.5181) | -0.266 (0.6911)

29. Secondary Outcome: Change From Baseline in CRP for Part 1
Description: Blood samples were collected at indicated time points for the assessment of CRP. Baseline was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value.
Time Frame: Baseline, Days 2, 4 and 7
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
mg/L
  Day 2 | -0.074 (0.1852) | 0.448 (0.7342) | 4.550 (3.8044) | 10.413 (10.7622) | 11.900 (6.1323) | 19.442 (1.9676)
  Day 4 | -0.101 (0.3839) | 0.098 (0.1480) | 0.748 (0.5974) | 2.430 (2.3835) | 2.362 (1.4852) | 3.760 (1.2465)
  Day 7 | 0.468 (1.3130) | 0.338 (0.3712) | 0.128 (0.3022) | 4.802 (9.2888) | 1.305 (0.8481) | 1.428 (1.0400)

30. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of GSK1795091 for Part 2
Description: Cmax assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of Adverse events (AEs) of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: PK Parameter Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

31. Secondary Outcome: Time of Occurrence of Cmax (Tmax) and Terminal Half Life (t1/2) of GSK1795091 for Part 2
Description: Tmax and t1/2 assessments were planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

32. Secondary Outcome: Partial Area Under the Concentration-time Curve to Time = t (AUC[0-t]), Area Under the Concentration-time Curve (AUC) From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of GSK1795091 for Part 2
Description: AUC (0-t) and AUC (0-inf) assessments were planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

33. Secondary Outcome: Area Under the Concentration-time Curve (AUC) Time Curve for a Dosing Interval (AUC[0-tau]), AUC (0-last) of GSK1795091 for Part 2
Description: AUC (0-tau) and AUC (0-last) assessments were planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

34. Secondary Outcome: Clearance (CL) of GSK1795091 for Part 2
Description: CL assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

35. Secondary Outcome: Volume of Distribution of GSK1795091 for Part 2
Description: Volume of distribution assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

36. Secondary Outcome: Accumulation Ratio of GSK1795091 for Part 2
Description: Accumulation ratio assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: PK Parameter Population. Data were not collected for part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

37. Secondary Outcome: Time Invariance of GSK1795091 for Part 2
Description: Time invariance assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Pre-dose, 5 minutes, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 144 hours post-dose
Population: as for outcome 30
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

38. Secondary Outcome: Percentage Fold Change of Concentration of Interleukin 6 (IL-6) From Baseline for Part 2
Description: IL-6 assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

39. Secondary Outcome: Percentage Fold Change of Concentration of TNF-alpha From Baseline for Part 2
Description: TNF-alpha assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

40. Secondary Outcome: Percentage Fold Change of Concentration of IFN-gamma From Baseline for Part 2
Description: IFN-gamma assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

41. Secondary Outcome: Percentage Fold Change of Concentration of IP-10 From Baseline for Part 2
Description: IP-10 assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. The data was not collected for Part 2 because no Par. were enrolled into this part of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

42. Secondary Outcome: Percentage Fold Change of Concentration of MCP-1 From Baseline for Part 2
Description: MCP-1 assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

43. Secondary Outcome: Percentage Fold Change of Concentration of GCSF From Baseline for Part 2
Description: GCSF assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

44. Secondary Outcome: Percentage Fold Change of Concentration of IL-1Ra From Baseline for Part 2
Description: IL-1Ra assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. The data was not collected for Part 2 because no Par. were enrolled into this part of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

45. Secondary Outcome: Percentage Fold Change of Concentration of IL-10 From Baseline for Part 2
Description: IL-10 assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 1, 2, 4, 8, 12, 16, 24, 48 and 144 hours
Population: PD Population. The data was not collected for Part 2 because no Par. were enrolled into this part of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

46. Secondary Outcome: Change From Baseline in WBC Differential for Part 2
Description: WBC differential assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline, 2, 24 and 144 hours
Population: All Subjects Population. Data was not collected for Part 2 as none of the participant was enrolled into Part 2 of the study.
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

47. Secondary Outcome: Number of Participants With Urinalysis Parameters Outside Reference Range for Part 2
Description: Urinalysis as part of safety assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

48. Secondary Outcome: Number of Participants With Hematology Parameters Outside Reference Range in Part 2
Description: Hematology as part of safety assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

49. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters Outside Reference Range in Part 2
Description: Clinical chemistry as part of safety assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

50. Secondary Outcome: Change From Baseline in CRP for Part 2
Description: CRP assessment was planned for Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline and Pre-dose, 1, 2, 4, 8, 12, 16, 24, and 48 hours post dose
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

51. Secondary Outcome: Change From Baseline in Body Temperature for Part 2
Description: Body temperature was planned to be measured in Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline and up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

52. Secondary Outcome: Change From Baseline in SBP and DBP for Part 2
Description: SBP and DBP was planned to be measured in Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline and up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

53. Secondary Outcome: Change From Baseline in Respiratory Rate for Part 2
Description: Respiratory rate was planned to be measured in Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline and up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

54. Secondary Outcome: Change From Baseline in Pulse Rate for Part 2
Description: Pulse rate was planned to be measured in Part 2 after IV dose administration to healthy participants 1 or 2 Weeks after the first dose. Baseline (Day 1) was taken as the mean of the planned pre-dose measurements. Change from Baseline was defined as difference between the post-Baseline visit value and the Baseline value. The data for Part 2 of the study was not collected as the study was discontinued by the Sponsor prior to its scheduled start due to participant in Part 1 experienced the late occurrence of AEs of unknown etiology.
Time Frame: Baseline and up to Day 7
Population: as for outcome 46
Arm/Group | All Participants in Part 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 102 days
Description: Non-serious AEs and SAE for All Subjects Population in Part 1 was reported. Non-serious AEs and SAE data was not collected for Part 2 as none of the participants were enrolled into Part 2 of the study.
Arm/Group | Part 1: Placebo | Part 1: GSK1795091 7 ng | Part 1: GSK1795091 21 ng | Part 1: GSK1795091 60 ng | Part 1: GSK1795091 Repeated 60 ng | Part 1: GSK1795091 100 ng | All Participants in Part 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 2/6 | 0/6 | 5/6 | 3/6 | 5/6 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=10) | Part 1: GSK1795091 7 ng (N=6) | Part 1: GSK1795091 21 ng (N=6) | Part 1: GSK1795091 60 ng (N=6) | Part 1: GSK1795091 Repeated 60 ng (N=6) | Part 1: GSK1795091 100 ng (N=6) | All Participants in Part 2 (N=0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02798978/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02798978/SAP_001.pdf